CLINICAL TRIAL: NCT05869357
Title: Safety of Cream Containing Sericin and Turmeric in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EC22010-20
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Safety Issues
MeSH Terms: interventions — Sericins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cream containing 2.5% sericin and 2%turmeric (Experimental): cream containing 2.5% sericin and 2%turmeric
  Interventions: Other: cream containing 2.5% sericin and 2%turmeric
- cream containing 5%sericin and 2%turmeric (Experimental): cream containing 5% sericin and 2%turmeric
  Interventions: Other: cream containing 5%sericin and 2%turmeric
- cream containing 10%sericin and 2%turmeric (Experimental): cream containing 10% sericin and 2%turmeric
  Interventions: Other: cream containing 10%sericin and 2%turmeric
- cream base (Experimental): cream base without sericin and tumeric
  Interventions: Other: cream base

INTERVENTIONS:
Other: cream containing 2.5% sericin and 2%turmeric — Sample is applied 2 times/day for 6 days. Then, use of the sample is stopped for 7 to 10 days. After that, sample is applied 2 times/day for 3days.
  Arms: cream containing 2.5% sericin and 2%turmeric
Other: cream containing 5%sericin and 2%turmeric — Sample is applied 2 times/day for 6 days. Then, use of the sample is stopped for 7 to 10 days. After that, sample is applied 2 times/day for 3days.
  Arms: cream containing 5%sericin and 2%turmeric
Other: cream containing 10%sericin and 2%turmeric — Sample is applied 2 times/day for 6 days. Then, use of the sample is stopped for 7 to 10 days. After that, sample is applied 2 times/day for 3days.
  Arms: cream containing 10%sericin and 2%turmeric
Other: cream base — Sample is applied 2 times/day for 6 days. Then, use of the sample is stopped for 7 to 10 days. After that, sample is applied 2 times/day for 3days.
  Arms: cream base

SUMMARY:
The object of this study was to evaluate safety of cream containing sericin and turmeric in healthy volunteers.

DETAILED DESCRIPTION:
There are 106 healthy volunteers in this study. Upper left arm is divided into 2 parts (2x2 cm) which are A and B area. Upper right arm is divided into 2 parts (2x2 cm) which are C and D area. Four area (A, B, C, and D) are randomized to receive cream containing 2.5% sericin and 2%turmeric, cream containing 5%sericin and 2%turmeric, cream containing 10%sericin and 2%turmeric, and cream base (Control group). Samples are applied 2 times/day for 6 days (Induction phase). Then, the volunteers will stop applying samples for 7 to 10 days (Free period). After that, Samples are applied 2 times/day for 3 days (Challenge phase). Erythema, melanin, humidity, transepidermal water loss, skin adverse reaction, and satisfaction are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* No skin diseases
* No allergy to sericin and turmeric
* No immunocompromised disease or using steroid for 2 weeks before participated in this study
* Willing to participate in this study

Exclusion Criteria:

* Uncontrolled disease, cancer, and heart disease
* Cannot follow the protocol
* Pregnancy and lactation
* Participated in other studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Erythema index | 19 days
  Measure by Cutometer. It represents inflammation. The value present in scale of erythema index (0 to 1000) (high value mean a worse outcome).
Melanin index | 19 days
  Measure by Cutometer. It represents post-inflammatory reaction. The value present in scale of melanin index (0 to 1000) (high value mean a worse outcome).

SECONDARY OUTCOMES:
Humidity index | 19 days
  Measure by Cutometer. It represents skin humidity. The value present in scale of humidity index (0 to 1000) (high value mean a better outcome).
Transepidermal water loss index | 19 days
  Measure by Cutometer. It represents skin water loss. The value present in scale of transepidermal water loss index (0 to 1000) (high value mean a worse outcome).
Skin reaction | 19 days
  Found or not found
Satisfaction of the volunteers | 19 days
  Measure by visual analogue scale (1 to 10 score means low satisfaction to high satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Pornanong Aramwit, Professor, Principal Investigator — Chulalongkorn University
Locations (1):
- Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn Unviersity, Bangkok, Thailand